CLINICAL TRIAL: NCT04958317
Title: The Effect of Exercise Timing on Postprandial Glycaemic Control: a Randomised Crossover Trial in Healthy Adults
Brief Title: Night Time Walking to Improve Glycaemic Control in Healthy Adults
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was planned for 2020, but Melbourne 2020 and 2021 lockdowns hindered the study.
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Barbara R. Cardoso, PhD, Monash University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Night Glucose response-walk
Record Dates: First submitted 2021-07-09; First posted 2021-07-12 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Postprandial Hyperglycemia; Insulin Resistance
Keywords: glucose tolerance; meal timing; insulin; postprandial; walking
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Who Masked: Investigator
Masking Description: This is a single masking study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early exercise (Placebo Comparator): Participants will exercise for 30 minutes prior to an evening meal
  Interventions: Other: Early exercise
- Late exercise (Experimental): Participants will exercise for 30 minutes after an evening meal
  Interventions: Other: Late exercise

INTERVENTIONS:
Other: Early exercise — Participants will exercise for 30 minutes prior to an evening meal.
  Arms: Early exercise
Other: Late exercise — Participants will exercise for 30 minutes after an evening meal.
  Arms: Late exercise

SUMMARY:
Randomised crossover trial to compare early vs late walking on postprandial glycaemic response at night time.

DETAILED DESCRIPTION:
In this crossover trial, eligible participants will be randomised to a 30-minute bout of physical activity (30 minute walk) either during the day or after an evening meal. The postprandial response to the evening meal will be analysed.

ELIGIBILITY:
Inclusion criteria

* Men and Women aged 18 to 65 years of age
* Waist circumference of <94cm and <80cm for Caucasian males and females, respectively
* Waist circumference of <90cm and <80 cm for Asian males and females, respectively
* Willingness to provide written informed consent and willingness to participate and comply with the study

Exclusion criteria

* Current or recent treatment (within 6 months) with medications that influence blood glucose
* Fasting blood glucose ≥ 7 mmol/L
* Individuals diagnosed with type 1 or type 2 diabetes mellitus, chronic gastrointestinal disorders (including inflammatory bowel disease and celiac) or any other condition deemed unstable
* Serious health conditions that may affect participation e.g. liver or thyroid dysfunction, recent major surgery
* Not able to walk for 30 mins at 5-5.5 km/hr
* Women planning pregnancy, pregnant or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Postprandial glucose | Three hour glucose iAUC will be calculated at nine time points (0, 15, 30, 45, 60, 90, 120, 150 and 180 mins) after beginning consumption of the test meal.
  Change in glucose incremental area under the curve (iAUC) in response to a meal challenge

SECONDARY OUTCOMES:
Postprandial insulin | Three hour insulin iAUC will be calculated at six time points (0, 30, 60, 90, 120 and 180 mins) after beginning consumption of the test meal.
  Change in insulin incremental area under the curve (iAUC) in response to a meal challenge

IPD SHARING:
Plan to Share IPD: No